CLINICAL TRIAL: NCT01869738
Title: MGuard™ Prime Stent System Clinical Trial in Patients With Acute ST Elevation Myocardial Infarction
Acronym: MASTER-II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment rate
Sponsor: InspireMD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMD-10
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: heart attack
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MGuard Prime (Experimental): MGuard Prime stent
  Interventions: Device: MGuard Prime
- Control (Active Comparator): (BMS/DES) Includes FDA approved bare metal or drug eluting stents, including ENDEAVOR, TAXUS Liberte, XIENCE Prime, PROMUS Element, ION, RESOLUTE, Driver, Vision, VeriFlex and Integrity.
  Interventions: Device: (BMS/DES)

INTERVENTIONS:
Device: MGuard Prime
  Arms: MGuard Prime
Device: (BMS/DES)
  Arms: Control

SUMMARY:
To evaluate the safety and efficacy of the MGuard™ Prime stent in the treatment of blocked arteries in coronary arteries in patients undergoing a stenting procedure due to having a heart attack. The MGuard Prime stent wil be compared to other FDA approved bare-metal (BMS) or drug-eluting (DES) coronary stents. The hypotheses are that (1) the MGuard Prime stent will achieve a higher rate of complete ST-segment resolution as seen on the post-procedure ECG as compared to the comparator stent, and will have a similar effect on the rate of all-cause death or recurrent target vessel myocardial infarction at 365 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is more than 18 years of age
* Subject is experiencing clinical symptoms consistent with acute myocardial infarction (AMI) of more than 30 minutes and less than 12 hours in duration.
* ST elevation more than 2 mm per lead in more than 2 contiguous leads is present in one ECG prior to consent.
* Subject agrees to all required follow-up procedures and visits.
* Subject or legal representative provides written, informed consent.
* The target lesion is a de novo lesion in a native coronary artery.
* Based on coronary anatomy, PCI is indicated for the culprit lesion with anticipated use of stenting.
* The reference vessel diameter (RVD) of the infarct lesion is 2.75 to 4.0 mm by visual assessment, assessed either at baseline (if direct stenting is planned), or after pre-dilatation or thrombus aspiration (if direct stenting is not planned).
* The entire lesion length requiring treatment is less than 24 mm (able to be covered by a single study stent), assessed either at baseline (if direct stenting is planned), or after pre-dilatation or thrombus aspiration (if direct stenting is not planned)
* TIMI flow of 2/3 is present prior to randomization (in case of baseline TIMI flow 0/1, blood flow must be restored).

Exclusion Criteria:

* Left bundle branch block (LBBB), paced rhythm, or other ECG abnormality interfering with assessment of ST-segment.
* Currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
* A previous coronary interventional procedure of any kind within 30 days prior to the procedure.
* Female patients of childbearing potential.
* Subject undergoing cardiopulmonary resuscitation (patients in whom cardiopulmonary resuscitation was successfully performed and in whom normal mental status was achieved, may be enrolled).
* Cardiogenic shock (SBP less than 80 mmHg for more than other hemodynamic support device for hypotension).
* The subject requires a staged procedure of the target vessel (including branches) within 12 months or of any non-target vessel within 7 days post-procedure.
* The target lesion requires treatment with a device other than PTCA prior to stent placement (such as, but not limited to excimer laser, rotational atherectomy, etc.). Manual thrombus aspiration may be used per operator discretion, but rheolytic thrombectomy is only permitted for procedural complications after randomization.
* Prior administration of thrombolytic therapy for the current admission
* Co-morbid condition(s) that could limit the subject's ability to participate in the trial or to comply with follow-up requirements, or impact the scientific integrity of the trial.
* Concurrent medical condition with a life expectancy of less than 12 months.
* History of cerebrovascular accident or transient ischemic attack within the last 6 months, or any permanent neurologic deficit
* Prior intracranial bleed at any time, or known intracranial pathology (e.g. tumor, arteriovenous malformation, or aneurysm).
* Active or recent site of major bleeding within 6 months.
* History of bleeding diathesis or coagulopathy or inability to accept blood transfusions.
* Known hypersensitivity or contraindication to either i) aspirin, or heparin and bivalirudin; or ii) clopidogrel , ticlopidine, prasugrel and ticagrelor; or iii) cobalt or nickel; or iv) contrast media, which cannot be adequately pre-medicated (prior anaphylaxis, however, is an absolute contraindication to enrollment).
* Known serum creatinine level more than 2.5 mg/dl, hemoglobin less than 10 g/dL or platelet count less than 150,000 for the present admission or within 7 days prior to index procedure, if available.
* Surgery planned or any other reason necessitating discontinuation of dual anti-platelet therapy (aspirin and an ADP antagonist) within 12 months
* Aortic dissection or mechanical complication of STEMI
* Unprotected left main stenosis more than 50%.
* Multi-vessel intervention required during the index procedure.
* Excessive tortuosity, calcification or diffuse distal disease
* A non-infarct lesion with stenosis more than 50% is present in the target vessel
* Target lesion is a bifurcation with a side branch more than 2.0 mm in diameter.
* Target lesion at the site of or within a vessel with a previously implanted stent
* Target lesion is within a bypass graft conduit, or can only be reached by passing the study stent through a bypass graft conduit
* In the Investigator's opinion the lesion/vessel is unsuitable for treatment with the study stent for any reason.
* The lesion requires use of atherectomy, thrombectomy (not including manual thrombus aspiration catheters), laser devices, or proximal or distal embolic protection devices prior to randomization.
* Aortic dissection or mechanical complication of STEMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
rate of complete ST-segment resolution within 60-90 minutes | 60-90 minutes post-procedure
The primary safety endpoint is a composite of all-cause death or recurrent target vessel myocardial infarction (TV re-MI) at 365 days post-procedure, powered to demonstrate non-inferiority of the MGuard™ Prime Stent compared to the control arm. | 365 days post-procedure

SECONDARY OUTCOMES:
Infarct size assessed by cardiac magnetic resonance imaging (MRI) | 5 days post-procedure
In-stent late lumen loss (LLL) | 13 months post-procedure

CONTACTS AND LOCATIONS:
Locations (56):
- United States (20):
  - Yale University School of Medicine, New Haven, Connecticut
  - Pepin Heart Hospital, Tampa, Florida
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Cardiology Associates of North Mississippi, Oxford, Mississippi
  - Valley Hospital, Ridgewood, New Jersey
  - Columbia University Medical Center, New York, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Elyria Memorial Hospital, Oberlin, Ohio
  - Northwest Ohio Cardiology, Toledo, Ohio
  - Holy Spirit Hospital, Camp Hill, Pennsylvania
  - Geisinger Clinic Cardiology, Danville, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - University of Virginia Health System, Charlottesville, Virginia
  - Winchester Medical Center, Winchester, Virginia
- ZNA Antwerpem, Antwerp, Belgium
- Czechia (2):
  - University hospital, Hradec Králové
  - Na Homolce Hospital, Prague
- North-Estonia Regional Hospital, Tallinn, Estonia
- Helsinki University Hospital, Helsinki, Finland
- France (5):
  - Hopital Henri Mondor, Créteil
  - Hopital Louis Pradel, Lyon
  - Institut Jacques Cartier, Massy
  - Hôpitaux GHI Le Raincy - Montfermeil, Montfermeil
  - Hôptal Européen Georges Pompidou, Paris
- Germany (5):
  - Charité Universitätsklinikum Berlin Campus Benjamin Franklin, Berlin
  - Charité Universitätsklinikum Berlin Campus Virchow, Berlin
  - Stadtische Kliniken München, Munich
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Universitat Ulm, Ulm
- Rabin Medical Center, Petah Tikva, Israel
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, AC
  - VU University Medical Center, Amsterdam
  - Academic Medical Center, Amsterdam
  - Albert Schweitzerziekenhuis, Dordrecht
- Poland (8):
  - Malopolskie Centrum Sercowo-Naczyniowe, Chrzanów
  - Polsko-Amerykańskie Kliniki Serca, Dąbrowa Górnicza
  - Górnośląskie Centrum Medyczne, Katowice
  - Krakowskie Centrum Kardiologii Inwazyjnej, Krakow
  - Szpital Uniwersyteckiw Krakowie, Krakow
  - John Paul II Hospital, Krakow
  - Katedra i Klinika Kardiologii Uniwersytetu Medycznego w Łodzi, Lodz
  - Klinika Kardiologii i Angiologii Interwencyjnej, Warsaw
- Spain (3):
  - Hospital Clinic, University of Barcelona, Barcelona
  - Bellvitge University Hospital, Barcelona
  - Hospital Universitario Madrid Montepríncipe, Madrid
- United Kingdom (5):
  - Bristol Heart Institute, Bristol
  - University Hospital of Wales, Cardiff
  - Golden Jubilee National Hospital, Glasgow
  - Leeds General Infirmary, Leeds
  - University Hospitals Southampton NHS Foundation Trust, Southampton